CLINICAL TRIAL: NCT04206657
Title: Pharmacokinetic Study of KHK7580 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Collaborators: Kyowa Kirin China Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 7580-202
Record Dates: First submitted 2019-12-18; First posted 2019-12-20 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Single dose administration of 1mg KHK7580 (Experimental)
  Interventions: Drug: 1mg KHK7580
- Single dose administration of 3mg KHK7580 (Experimental)
  Interventions: Drug: 3mg KHK7580
- Single dose administration of 6mg KHK7580 (Experimental)
  Interventions: Drug: 6mg KHK7580
- Single dose administration of 12mg KHK7580 (Experimental)
  Interventions: Drug: 12mg KHK7580
- Multiple dose administration of 6mg KHK7580 for 8days (Experimental)
  Interventions: Drug: 6mg KHK7580 for 8days

INTERVENTIONS:
Drug: 1mg KHK7580 — Single oral dose administration of 1mg KHK7580
  Arms: Single dose administration of 1mg KHK7580
Drug: 3mg KHK7580 — Single oral dose administration of 3mg KHK7580
  Arms: Single dose administration of 3mg KHK7580
Drug: 6mg KHK7580 — Single oral dose administration of 6mg KHK7580
  Arms: Single dose administration of 6mg KHK7580
Drug: 12mg KHK7580 — Single oral dose administration of 12mg KHK7580
  Arms: Single dose administration of 12mg KHK7580
Drug: 6mg KHK7580 for 8days — multiple oral dose administration of 6mg KHK7580 for 8days
  Arms: Multiple dose administration of 6mg KHK7580 for 8days

SUMMARY:
The primary objective is to evaluate the pharmacokinetic profile of KHK7580 in Chinese healthy adult volunteers. The secondary objective is to evaluate its safety and pharmacodynamics.

ELIGIBILITY:
Inclusion Criteria:

1. Personally submitted written voluntary informed consent to participate in the study;
2. Chinese adult ≥20 and <40 years of age at informed consent;
3. BMI ≥18.5 kg/m2 and <25.0 kg/m2 at screening.

Exclusion Criteria:

Subjects must be excluded from the study if they meet any of the following criteria:

1. Subjects with present illness requiring treatment;
2. Subjects in whom the serum Ca concentration, as measured at pretreatment (screening and Day -1) blood chemistry examination, is below the lower limit of the in-house reference value;
3. Subjects in whom a clinically significant abnormality in the crystalline lens is noted at a pre-study ophthalmological examination;
4. Subjects with urinary tract lithiasis or its past history;
5. Subjects with convulsive seizure or its past history;
6. Subjects with digestive system disorder (peptic ulcer, reflux esophagitis, etc.) or its past history (in this regard, however, a past history of appendicitis is acceptable);
7. Subjects with mental disorder or its past history;
8. Subjects who have alcohol/drug dependence or tested positive for any of the drug abuse test items;
9. Subjects with symptomatic allergy disease;
10. Subjects with drug allergy or its past history;
11. Subjects with a past history or family history of congestive heart failure, hypokalemia, or long QT syndrome; Protocol Number: 7580-202 (ver. 1.2) Date: 25 April, 2019 CONFIDENTIAL 7
12. Subjects in whom a 12-lead ECG tracing before initiation of study drug administration showed, in the judgment of the investigator or subinvestigator, a clinically significant abnormality or an electrocardiographic waveform shape unfit for QT interval measurement;
13. Subjects who tested positive for any of the infection test items;
14. Subjects who have used any drugs (including over-the-counter drugs, external preparations, vitamin preparations, and herbal preparations) within 2 weeks before initiation of study drug administration;
15. Subjects who have smoked a cigarette or used a treatment aid to smoking cessation (including nicotine-containing product chewing/ingestion and nicotine-containing patches) within 2 weeks before initiation of the study drug administration;
16. Subjects who have participated in a clinical study of a drug and practically received the drug within 4 months before initiation of the study drug administration;
17. Subjects who, within 3 months before initiation of the study drug administration, have been hospitalized, undergone surgery, or undergone collection of at least 200 mL of blood (including blood donation and blood component donation);
18. Subjects who did not consent to use an effective contraceptive (e.g., use of condoms) alone or in combination between the day of hospitalization and 3 months after the end of the study drug administration;
19. Pregnant, lactating, possibly pregnant subjects/women (subjects/women of childbearing potential with positive pregnancy test at screening or Day -1, or with negative pregnancy test at screening and Day -1 not using any contraceptive methods), or unwilling to use adequate contraception according to the physician's instructions. Amenorrhea for ≥12 months after the last menstrual period without an alternative medical cause is considered as non-childbearing potential;
20. Prior exposure to KHK7580;
21. Other conditions unfit for participation in this study at the discretion of the investigator or subinvestigator.

Ages: 20 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2021-06-17 (Actual); Study Completion 2021-06-17 (Actual)

PRIMARY OUTCOMES:
Plasma KHK7580 concentration at each time point | pre-dose, 0.25, 0.5,1,2,3,4,6,8,12,24,36,48,72 hours post-dose for single dose cohort; pre-dose, 0.25, 0.5,1,2,3,4,8,12,16 hours post dose of Day -1 and pre-dose, 2,4,8,12,16,24,36,48,72,96 hours post-dose of Day 8 for multiple dose cohort
Time to Reach Maximum Observed Plasma Concentration (Tmax) of KHK7580 | pre-dose, 0.25, 0.5,1,2,3,4,6,8,12,24,36,48,72 hours post-dose for single dose cohort; pre-dose, 0.25, 0.5,1,2,3,4,8,12,16 hours post dose of Day -1 and pre-dose, 2,4,8,12,16,24,36,48,72,96 hours post-dose of Day 8 for multiple dose cohort
Maximum Observed Plasma Concentration (Cmax) of KHK7580 | pre-dose, 0.25, 0.5,1,2,3,4,6,8,12,24,36,48,72 hours post-dose for single dose cohort; pre-dose, 0.25, 0.5,1,2,3,4,8,12,16 hours post dose of Day -1 and pre-dose, 2,4,8,12,16,24,36,48,72,96 hours post-dose of Day 8 for multiple dose cohort
Area under the plasma concentration-time curve from time 0 to the time of last quantifiable concentration (AUC0-t) of KHK7580 | pre-dose, 0.25, 0.5,1,2,3,4,6,8,12,24,36,48,72 hours post-dose for single dose cohort; pre-dose, 0.25, 0.5,1,2,3,4,8,12,16 hours post dose of Day -1 and pre-dose, 2,4,8,12,16,24,36,48,72,96 hours post-dose of Day 8 for multiple dose cohort
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of KHK7580 | pre-dose, 0.25, 0.5,1,2,3,4,6,8,12,24,36,48,72 hours post-dose for single dose cohort; pre-dose, 0.25, 0.5,1,2,3,4,8,12,16 hours post dose of Day -1 and pre-dose, 2,4,8,12,16,24,36,48,72,96 hours post-dose of Day 8 for multiple dose cohort
Plasma Half-Life (t1/2) of KHK7580 | pre-dose, 0.25, 0.5,1,2,3,4,6,8,12,24,36,48,72 hours post-dose for single dose cohort; pre-dose, 0.25, 0.5,1,2,3,4,8,12,16 hours post dose of Day -1 and pre-dose, 2,4,8,12,16,24,36,48,72,96 hours post-dose of Day 8 for multiple dose cohort
Apparent systemic clearance (CL/F) of KHK7580 | pre-dose, 0.25, 0.5,1,2,3,4,6,8,12,24,36,48,72 hours post-dose for single dose cohort; pre-dose, 0.25, 0.5,1,2,3,4,8,12,16 hours post dose of Day -1 and pre-dose, 2,4,8,12,16,24,36,48,72,96 hours post-dose of Day 8 for multiple dose cohort

SECONDARY OUTCOMES:
Incidence of treatment emergent adverse events (TEAEs) | Dosing to study completion
QTcF | [Single dose] baseline to Day 4; [Multiple dose] baseline to Day 12
QTcB | [Single dose] baseline to Day 4; [Multiple dose] baseline to Day 12
intact PTH level | [Single dose] baseline to Day 4; [Multiple dose] baseline to Day 12
serum P level | [Single dose] baseline to Day 4; [Multiple dose] baseline to Day 12

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided